CLINICAL TRIAL: NCT03403751
Title: Phase 3 Randomized, Double-blind Study to Evaluate the Safety and Efficacy of Reltecimod as Compared to Placebo in Addition to Standard of Care in Patients With Sepsis-associated Acute Kidney Injury (SA-AKI)
Brief Title: Phase 3 Study of Reltecimod vs Placebo in Patients With Sepsis-associated Acute Kidney Injury
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Very slow enrollment of target patient population
Sponsor: Atox Bio Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATB-203
Record Dates: First submitted 2018-01-06; First posted 2018-01-19 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Acute Kidney Injury; Peritonitis; Necrotizing Soft Tissue Infection
Keywords: Abdominal sepsis; AKI; NSTI
MeSH Terms: conditions — Acute Kidney Injury; Peritonitis; Intraabdominal Infections | interventions — AB103; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of study drug (Reltecimod) and placebo (normal saline)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor personnel and clinical research associates (CRAs) will also be blinded to study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reltecimod 0.5 mg/kg (Experimental): Single IV infusion of Reltecimod 0.5 mg/kg
  Interventions: Drug: Reltecimod 0.5 mg/kg
- Placebo (Placebo Comparator): Single IV infusion of 0.9% Sodium Chloride Injection (Normal Saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reltecimod 0.5 mg/kg — Single IV infusion of 0.5 mg/kg Reltecimod (at a concentration of 1 mg/mL) over approximately 10 minutes
  Other Names: AB103 0.5 mg/kg
  Arms: Reltecimod 0.5 mg/kg
Drug: Placebo — Single IV infusion of 0.5 mL/kg of 0.9% saline (volume equivalent to Reltecimod dosing schema) over approximately 10 minutes
  Other Names: 0.9% Sodium Chloride Injection (Normal saline)
  Arms: Placebo

SUMMARY:
Phase 3 multicenter study to be conducted in up to 90 qualified participating sites globally to assess the efficacy and safety of Reltecimod vs placebo in patients with sepsis-associated Stage 2/3 AKI.

DETAILED DESCRIPTION:
Phase 3 randomized, placebo controlled study assessing the efficacy (complete recovery from AKI) and safety of Reltecimod in patients with suspected or confirmed abdominal sepsis (planned or completed surgical (laparotomy or laparoscopy) or interventional radiologic procedures for control of underlying abdominal infection within 24 hours of evaluation by medical personnel) or patients with surgically confirmed necrotizing soft tissue infection (NSTI), requiring intensive care unit (ICU) or step down unit admission and in whom the diagnosis of Stage 2/3 acute kidney injury (AKI; as defined by Kidney Disease Improving Global Outcomes (KDIGO) criteria) is established at initial presentation for medical evaluation or up to 48 hours from the suspected diagnosis of abdominal sepsis or from surgically confirmed diagnosis of NSTI.

ELIGIBILITY:
Inclusion Criteria:

1. Has either suspected or documented diagnosis of abdominal sepsis requiring treatment with parenteral antibiotics and planned or completed surgical (laparotomy or laparoscopy) or interventional radiologic procedures within 24 hours of evaluation by medical personnel. Recommended surgical or interventional radiologic procedures be performed with 12 hours of evaluation by medical personnel.
2. Initial diagnosis of AKI Stage 2 or 3 according to KDIGO AKI criteria established either upon presentation to medical care in those patients with suspected abdominal sepsis or in those patients in whom the initial diagnosis of AKI is established during the 48 hour period from the suspected diagnosis of abdominal sepsis.
3. Study medication must be administered within 6 hours of confirmation of onset of Stage 2 or 3 AKI as established at the study site, under the following criteria:

   * After the decision is made by the attending surgeon at the study site for a surgical or interventional radiology procedure for the abdominal infection OR
   * After confirmed diagnosis of abdominal infection has been established by a surgical or interventional radiology procedure

Exclusion Criteria:

1. Has known prior history of chronic kidney disease (CKD( with a documented estimated GFR (eGFR) < 30 mL/min

   • Exception: Patients with history of CKD but no available prior eGFR who have documented normal kidney size on ultrasound or computed tomography evaluation (performed within 90 days of screening) will be eligible
2. Patients receiving renal replacment therapy (RRT) for CKD
3. . Previously diagnosed with documented AKI in the last 30 days
4. Documented primary glomerular disease or toxic tubulo-interstitial nephritis at the time of AKI diagnosis
5. Patient is not expected to survive throughout 28 days of study due to significant underlying medical condition
6. Any concurrent medical condition, which in the opinion of the Investigator, may compromise the safety of the patient or the objectives of the study or the patient will not benefit from treatment such as:

   * Congestive heart failure (CHF) {New York Heart Association (NYHA) class III-IV}
   * Severe chronic obstructive pulmonary disease (COPD) {GOLD - Global Initiative for Chronic Obstructive Lung Disease - stage IV. or chronic hypoxemia)
   * Liver dysfunction {Childs-Pugh class C}
   * Primary or acquired immunodeficiency or immunosuppression due to treatment with immunosuppressive medications
   * Known HIV infection with CD4 count < 200 cells/mm3 or < 14% of all lymphocytes
   * Neutropenia < 1,000 cells/mm3 not due to the underlying infection
   * Receiving or about to receive chemotherapy or biologic anti-cancer treatment,
   * Hematological and lymphatic malignancies in the last 5 years
7. Patient has acute pancreatitis with no established source of infection, uncomplicated appendicitis, or cholangitis or cholecystitis without peritonitis;
8. Pregnant or lactating women
9. Concurrent or previous enrollment in a clinical trial involving investigational drug or a medical device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azra Bihorac, MD, Principal Investigator — University of Florida Health
Locations (56):
- United States (40):
  - Maricopa Medical Center, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - University of California, Davis Medical Center, Sacramento, California
  - UCSD Medical Center, San Diego, California
  - Harbor-UCLA Medical Center, Torrance, California
  - UCH-Memorial Health System, Colorado Springs, Colorado
  - University of Colorado Hospital, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - LSU Health Science Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Capital Health System, Inc., Trenton, New Jersey
  - Erie County Medical Center-Affliate of SUNYat Buffalo, Buffalo, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati Medical Center (UCMC), Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - The Pennsylvania State University and The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Trauma Center at PENN, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MUSC, Charleston, South Carolina
  - John Peter Smith Health Network, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- France (16):
  - Hopital Victor Dupouy, Argenteuil
  - CHRU la Cavale Blanche, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHD Vendee, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - Robert Salengro Hopital-CHRU Lille, Lille
  - CHU de Limoges, Limoges
  - CHU Lyon Sud, Lyon
  - Hopital Edouard Herriot, Lyon
  - Hopital Saint Eloi, Montpellier
  - CHU de Nante Hotel-Dieu, Nantes
  - CHU Nimes, Nîmes
  - Hopital Cochin, Paris
  - CHU Rennes, Rennes
  - Nouvel Hopital Civil, Strasbourg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Reltecimod 0.5 mg/kg: Single IV infusion of 0.5 mg/kg Reltecimod (at a concentration of 1 mg/mL)
- Placebo: Single IV infusion of 0.5 mL/kg of 0.9% sodium chloride (volume equivalent with Reltecimod dosing schema)
Period: Overall Study
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Started | 28 | 30
Completed | 21 | 22
Not Completed | 7 | 8
Not completed — Death | 5 | 6
Not completed — Discontinuation (includes missing from Day 29) | 2 | 2

BASELINE CHARACTERISTICS:
Population: This analysis population included all randomized patients who were exposed to study drug (reltecimod or placebo) and who had a suspected or confirmed diagnosis of abdominal sepsis or confirmed NSTI and Stage 2 or Stage 3 AKI, with patients analyzed according to the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reltecimod 0.5 mg/kg | Placebo | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (14.6) | 61.8 (13.6) | 61.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 12 | 15 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 23 | 29 | 52
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 23 | 22 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (6.9) | 32.3 (12.2) | 31.4 (9.9)
Disease Category [Count of Participants; unit: Participants]
  Abdominal Infection | 27 | 29 | 56
  Necrotizing Soft Tissue Infection (NSTI) | 1 | 1 | 2
Comorbidities [Count of Participants; unit: Participants]
  Diabetes | 11 | 6 | 17
  Cardiovascular Disease | 7 | 6 | 13
  Smoker | 1 | 5 | 6
  Alcohol Abuse | 1 | 2 | 3
Modified Sequential Organ Failure Assessment (mSOFA) Score [Mean (Standard Deviation); unit: score on a scale] — Modified Sequential Organ Failure Assessment (mSOFA) total scores range from 0 to 20, with higher scores reflecting a worse clinical status or outcome. An mSOFA total score of 0 or 1 reflects resolution of organ dysfunction/failure.
  score on a scale | 4.9 (2.3) | 5.4 (3.1) | 5.1 (2.8)
Acute Physiology and Chronic Health Evaluation (APACHE) Score [Mean (Standard Deviation); unit: score on a scale] — The Acute Physiology and Chronic Health Evaluation (APACHE) Score is a severity of illness classification system. It is determined within 24 hours of admission of a patient to an intensive care unit (ICU): an integer score from 0 to 71 is computed based on several measurements (physiologic variables, age, chronic health status).
  Higher scores correspond to more severe disease and a greater risk of death.
  score on a scale | 17.1 (8.5) | 16.4 (7.9) | 16.7 (8.2)
Sepsis Presentation [Count of Participants; unit: Participants]
  Cardiovascular Organ Failure | 12 | 17 | 29
  Respiratory Organ Failure | 2 | 3 | 5
Acute Kidney Injury (AKI) Presentation [Count of Participants; unit: Participants]
  Stage 2 AKI | 20 | 25 | 45
  Stage 3 AKI | 8 | 5 | 13
Acuity of AKI [Count of Participants; unit: Participants]
  AKI diagnosed at time of diagnosis of infection | 17 | 12 | 29
  AKI diagnosed during the 48h following diagnosis of infection | 11 | 18 | 29

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Durable Loss of Renal Function at Day 28
Description: Freedom from durable loss of renal function at Day 28 required all of the following 3 components: alive at Day 28, free of dialysis at Day 28, and less than 37% loss of estimated glomerular filtration rate (eGFR) at Day 28 from patient reference eGFR (measured by Modification of Diet in Renal Disease [MDRD] formula).
Time Frame: 28 Days
Population: This analysis population (modified intent-to-treat [mITT]) included all randomized patients who were exposed to study drug (reltecimod or placebo) and who had a suspected or confirmed diagnosis of abdominal sepsis or confirmed necrotizing soft tissue infection (NSTI) and Stage 2 or Stage 3 AKI, with patients analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
Participants | 20 | 23
Statistical Analysis 1: Comparison: Reltecimod 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.649, Chi-squared

2. Primary Outcome: Serious Adverse Events (SAEs)
Description: Number of patients experiencing at least one SAE
Time Frame: 28 Days
Population: This analysis population (As Treated/Safety Analysis Set) included all randomized patients who were exposed to study drug (reltecimod or placebo), with patients analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
Participants | 12 | 13

3. Primary Outcome: Adverse Events (AEs)
Description: The number of patients experiencing at least one AE.
Time Frame: 28 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
Participants | 15 | 24

4. Secondary Outcome: Freedom From Durable Loss of Renal Function at Day 14
Description: Freedom from durable loss of renal function at Day 14 required all of the following 3 components: alive at Day 14, free of dialysis at Day 14, and less than 37% loss of estimated glomerular filtration rate (eGFR) at Day 14 from patient reference eGFR (measured by Modification of Diet in Renal Disease [MDRD] formula).
Time Frame: 14 Days
Population: This analysis population (modified intent-to-treat [mITT]) included all randomized patients who were exposed to study drug (reltecimod or placebo) and who had a suspected or confirmed diagnosis of abdominal sepsis or confirmed NSTI and Stage 2 or Stage 3 AKI, with patients analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
Participants | 20 | 22
Statistical Analysis 1: Comparison: Reltecimod 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.871, Chi-squared

5. Secondary Outcome: Intensive Care Unit (ICU)-Free Days
Description: ICU-free days refers to the number of days a patient did not spend time in the ICU through Day 28.
Time Frame: 28 Days
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
days | 24.0 [0 to 28] | 21.0 [0 to 28]
Statistical Analysis 1: Comparison: Reltecimod 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.420, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Ventilator-free Days
Description: Ventilator-free days refers to the number of days a patient was not on a ventilator through Day 28.
Time Frame: 28 Days
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
days | 26.5 [0 to 28] | 26.0 [0 to 28]
Statistical Analysis 1: Comparison: Reltecimod 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.448, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Vasopressor-free Days
Description: Vasopressor-free days refers to the number of days a patient did not receive a vasopressor through Day 28.
Time Frame: 28 Days
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
days | 27.5 [0 to 28] | 26.5 [0 to 28]
Statistical Analysis 1: Comparison: Reltecimod 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.579, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Hospital Days
Description: Hospital days refers to the number of days a patient spent time in the hospital.
Time Frame: 90 Days
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
days | 9.0 [2 to 61] | 13.0 [1 to 60]
Statistical Analysis 1: Comparison: Reltecimod 0.5 mg/kg vs Placebo; Test type: Superiority; p = 0.227, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Cumulative Number of Deaths
Description: The number of deaths occurring through Day 90
Time Frame: 90 Days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
Participants | 5 | 6

10. Secondary Outcome: Secondary Infections
Description: Number of patients experiencing at least one secondary infection
Time Frame: 28 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
Number analyzed (Participants) | 28 | 30
Participants | 4 | 10

11. Secondary Outcome: ICU-free Days by Day 14 Modified Sequential Organ Failure Assessment (mSOFA) Category
Description: The number of days a patient did not spend in the ICU through Day 28, by mSOFA category (mSOFA total score of 1 or less; mSOFA total score of 2 or more). Modified Sequential Organ Failure Assessment (mSOFA) total scores range from 0 to 20, with higher scores reflecting a worse clinical status or outcome. An mSOFA total score of 0 or 1 reflects resolution of organ dysfunction/failure.
Time Frame: 28 Days
Population: This analysis population (modified intent-to-treat [mITT]) included all randomized patients who were exposed to study drug (reltecimod or placebo) and who had a suspected or confirmed diagnosis of abdominal sepsis or confirmed NSTI and Stage 2 or Stage 3 AKI, with patients analyzed according to the treatment actually received. Only patients with available mSOFA data are included in the analysis.
Measure: Median (Full Range); unit: days
Groups:
- Day 14 mSOFA <= 1: mSOFA total score on Day 14 of 0 or 1
- Day 14 mSOFA >= 2: mSOFA total score on Day 14 of at least 2
Arm/Group | Day 14 mSOFA <= 1 | Day 14 mSOFA >= 2
Number analyzed (Participants) | 26 | 10
days | 24.0 [5 to 28] | 4.0 [0 to 26]
Statistical Analysis 1: Comparison: Day 14 mSOFA <= 1 vs Day 14 mSOFA >= 2; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Ventilator-free Days by Day 14 mSOFA Category
Description: The number of days a patient was not on a ventilator through Day 28, by mSOFA category
Time Frame: 28 Days
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | Day 14 mSOFA <= 1 | Day 14 mSOFA >= 2
Number analyzed (Participants) | 26 | 10
days | 27.0 [8 to 28] | 17.0 [1 to 28]
Statistical Analysis 1: Comparison: Day 14 mSOFA <= 1 vs Day 14 mSOFA >= 2; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Vasopressor-free Days by Day 14 mSOFA Category
Description: The number of days a patient was not receiving a vasopressor through Day 28, by mSOFA category
Time Frame: 28 Days
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | Day 14 mSOFA <= 1 | Day 14 mSOFA >= 2
Number analyzed (Participants) | 26 | 10
days | 28.0 [24 to 28] | 18.0 [0 to 28]
Statistical Analysis 1: Comparison: Day 14 mSOFA <= 1 vs Day 14 mSOFA >= 2; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Hospital Days by Day 14 mSOFA Category
Description: The number of days a patient was in the hospital.
Time Frame: 90 Days
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | Day 14 mSOFA <= 1 | Day 14 mSOFA >= 2
Number analyzed (Participants) | 26 | 10
days | 13.0 [4 to 48] | 23.5 [9 to 61]
Statistical Analysis 1: Comparison: Day 14 mSOFA <= 1 vs Day 14 mSOFA >= 2; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Hospital Discharge Location by Day 14 mSOFA Category
Description: Number of patients with more favorable discharge location (home or rehabilitation facility) or less favorable discharge location (skilled nursing facility, another acute care facility, death, other) among patients alive at Day 14.
Time Frame: 90 Days
Population: This analysis population (modified intent-to-treat [mITT]) included all randomized patients who were exposed to study drug (reltecimod or placebo) and who had a suspected or confirmed diagnosis of abdominal sepsis or confirmed NSTI and Stage 2 or Stage 3 AKI, with patients analyzed according to the treatment actually received. Only patients alive at Day 14 with available data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Day 14 mSOFA <= 1 | Day 14 mSOFA >= 2
Number analyzed (Participants) | 38 | 12
Participants
  More Favorable Discharge Location | 28 | 4
  Less Favorable Discharge Location | 10 | 8

16. Other Pre Specified Outcome: Cumulative Mortality by Day 14 mSOFA Category
Description: Percentage of patients who died through Day 90 using life table analysis
Time Frame: 90 Days
Population: This analysis population (modified intent-to-treat [mITT]) included all randomized patients who were exposed to study drug (reltecimod or placebo) and who had a suspected or confirmed diagnosis of abdominal sepsis or confirmed NSTI and Stage 2 or Stage 3 AKI, with patients analyzed according to the treatment actually received. Only patients with a screening mSOFA >= 3 are included in the analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Day 14 mSOFA <= 1 | Day 14 mSOFA >= 2
Number analyzed (Participants) | 26 | 10
percentage of patients | 0 | 31.4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) reported here were collected from study drug administration through the Day 29 visit (28 days after study drug dosing).
Description: Safety data obtained during study visits associated with Study Days 1, 2, 3, 7, 10, 14, 21, and 28 were systematically assessed throughout the study. In addition, data from spontaneously reported AEs were included in safety assessments.
Arm/Group | Reltecimod 0.5 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 5/28 | 6/30
Serious Adverse Events (participants affected / at risk) | 12/28 | 13/30
Other Adverse Events (participants affected / at risk) | 7/28 | 8/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reltecimod 0.5 mg/kg (N=28) | Placebo (N=30)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Organ failure (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal wall infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urethral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (2)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reltecimod 0.5 mg/kg (N=28) | Placebo (N=30)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT03403751/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT03403751/SAP_001.pdf